CLINICAL TRIAL: NCT01702506
Title: Phase 1 Three Period Crossover Study To Evaluate The Effect Of Food And Antacids On The Pharmacokinetics, Safety & Tolerability Of PF-299,804 In Healthy Volunteers Who Have Received PF-299,804
Brief Title: Evaluation Of The Potential Effect That The Administration Of Food Or Antacid Medication May Have In The Oral Absorption Of Dacomitinib (PF-00299804)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A7471015
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Healthy Volunteers
Keywords: Dacomitinib; PF-00299804; fed; fasted; antacid; relative Bioavailability
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fasted (Experimental): Dacomitinib administered under fasted conditions
  Interventions: Drug: dacomitinib fasted
- Fed (Experimental): Dacomitinib administered under fed conditions
  Interventions: Drug: dacomitinib fed
- Antacid (Experimental): Dacomitinib administered under antacid treatment
  Interventions: Drug: dacomitinib+antacid

INTERVENTIONS:
Drug: dacomitinib fasted — Overnight fasted subjects will receive a single 45 mg dose of dacomitinib
  Arms: Fasted
Drug: dacomitinib fed — Subjects will receive a single 45 mg dose of dacomitinib with a high calorie high fat meal
  Arms: Fed
Drug: dacomitinib+antacid — Subjects will receive a single 45 mg dose of dacomitinib when there are treated with rabeprazole
  Arms: Antacid

SUMMARY:
Evaluation of the potential effect that the administration of food or antacid medication may have in the oral absorption of dacomitinib relative to the administration of dacomitinib in absence of food or antacid medication

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects including males between the ages of 18 and 55 years. Females of non childbearing potential .
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject.

Exclusion Criteria:

* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or the appropriate time based on the elimination characteristics of the study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 2 weeks
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8). For dacomitinib and PF-05199265
Maximum Observed Plasma Concentration (Cmax) | 2 weeks
  For dacomitinib and PF-05199265

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] | 2 weeks
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t).For dacomitinib and PF-05199265
Area under the Concentration-Time Curve (AUC) | 3 days
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. For dacomitinib and PF-05199265
Apparent Oral Clearance (CL/F) | 2 weeks
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. For dacomitinib
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 2 weeks
  For dacomitinib and PF-05199265
Apparent Volume of Distribution (Vz/F) | 2 weeks
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed. For dacomitinib
Plasma Decay Half-Life (t1/2) | 2 weeks
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. For dacomitinib

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- [Derived] Ruiz-Garcia A, Masters JC, Mendes da Costa L, LaBadie RR, Liang Y, Ni G, Ellery CA, Boutros T, Goldberg Z, Bello CL. Effect of food or proton pump inhibitor treatment on the bioavailability of dacomitinib in healthy volunteers. J Clin Pharmacol. 2016 Feb;56(2):223-30. doi: 10.1002/jcph.588. Epub 2015 Oct 9. PMID 26179237
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471015&StudyName=Evaluation%20Of%20The%20Potential%20Effect%20That%20The%20Administration%20Of%20Food%20Or%20Antacid%20Medication%20May%20Have%20In%20The%20Oral%20Absorption%20Of%20Dacomitini